CLINICAL TRIAL: NCT06828029
Title: The Effect of Problem-Solving Approach Training on Professional Readiness Perception in Newly Graduated Nurses
Brief Title: Problem-Solving Approach Training on Professional Readiness Perception
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Seda Tugba Baykara Mat, Asst. Prof., University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: The Effect of Problem-Solving
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-01

CONDITIONS: Problem-solving
Keywords: Problem-Solving; Professional Readiness; Newly Graduated Nurses

STUDY DESIGN:
Intervention Model Description: The problem-solving training consists of five modules, blending theory and practice. Module 1 covers the basics of problem-solving, including key steps like identification, analysis, and evaluation, with group activities for hands-on practice. Module 2 focuses on creative techniques, such as brainstorming and mind mapping, to develop innovative solutions. Module 3 teaches decision-making and prioritization, using tools like SWOT analysis and decision trees, with applied exercises. Module 4 emphasizes teamwork and communication, highlighting conflict resolution and effective collaboration through team-based problem-solving activities. Module 5 integrates all techniques, applying them to real-life scenarios, particularly clinical cases, with group discussions and solution evaluations. The training incorporates interactive learning, simulations, and structured feedback, aiming to enhance problem-solving and leadership skills. Evaluation includes self-assessment and performance observation
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the experimental group who started working at the hospital (Experimental): Problem solving training was applied to the experimental group.
  Interventions: Behavioral: Problem-Solving
- control grubu (No Intervention): No training was provided.

INTERVENTIONS:
Behavioral: Problem-Solving — The problem-solving training consists of five modules, blending theory and practice. Module 1 covers the basics of problem-solving, including key steps like identification, analysis, and evaluation, with group activities for hands-on practice. Module 2 focuses on creative techniques, such as brainstorming and mind mapping, to develop innovative solutions. Module 3 teaches decision-making and prioritization, using tools like SWOT analysis and decision trees, with applied exercises. Module 4 emphasizes teamwork and communication, highlighting conflict resolution and effective collaboration through team-based problem-solving activities. Module 5 integrates all techniques, applying them to real-life scenarios, particularly clinical cases, with group discussions and solution evaluations. The training incorporates interactive learning, simulations, and structured feedback, aiming to enhance problem-solving and leadership skills. Evaluation includes self-assessment and performance observation
  Arms: the experimental group who started working at the hospital

SUMMARY:
The aim of this study is to examine the effect of problem-solving approach training on the professional readiness perception of newly hired nurses. Nursing practices are dynamic and require strong problem-solving abilities. In this context, the study will explore how the support provided through education during the transition period for new graduate nurses influences their perception of professional competence.

The hypothesis of the study is that problem-solving approach training will enhance the professional readiness perception of newly hired nurses. It is anticipated that the training will improve the nurses' professional knowledge and skills, equipping them to better handle the clinical challenges they will encounter.

The study is planned to take place between February and June 2025 at Zoom platform. The population of the study consists of newly hired nurses, and a sample size calculation has been performed using power analysis. Effect size (Cohen's d): An effect size of 0.5 (moderate effect) has been assumed for this study. Alpha level (α): A Type I error rate of 0.05 is used. Power (1 - β): A power of 0.90 (90%) has been targeted.

Using these parameters and the G*Power software, the sample size is calculated to be approximately 64 participants per group. Therefore, the target is to recruit at least 128 participants for the study.

Participants will be randomly assigned to experimental and control groups. The experimental group will receive online and interactive problem-solving approach training. Participants in the experimental group will be supported with problem-solving-based training modules, focusing on decision-making skills related to nursing practice throughout the training process. The control group will not receive any training. After the training, both groups' professional readiness perceptions will be assessed using the previously determined Personal Information Form and Professional Readiness Scale.

The data collected in the study will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 software. Kolmogorov-Smirnov test will be used to determine whether the data follows a normal distribution. If p > 0.05, the data will be considered to follow a normal distribution. If p < 0.05, the data will be considered not normally distributed, and skewness and kurtosis values will be examined. For repeated measures, if the data is normally distributed, repeated measures ANOVA will be used; if the data is not normally distributed, Friedman's test will be applied. Descriptive statistics will first be used to summarize the general characteristics of the data, and the means and distributions of pre-test and post-test scores will be determined. To evaluate the effect of the training intervention, paired samples t-test will be applied to assess the differences between pre-test and post-test scores within the same group. This analysis will be used to measure the effect of the training program on time management and procrastination behaviors. Additionally, effect size (e.g., Cohen's d) will be calculated to evaluate the magnitude and significance of the training intervention's effect. Analysis of variance (ANOVA) will be used to determine whether there are significant differences between the groups, depending on the study's needs.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Working for a maximum of 6 months
* Graduated from the Department of Nursing
* To know and understand Turkish at an adequate level
* Voluntary participation
* Access to online education platforms
* Participated in at least 4 out of 5 weekly trainings

Exclusion Criteria:

* Department/school change
* The student requests to leave the study
* Continuing formal education
* Not working at the hospital

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Professional Readiness | 5 months
  The scale developed by Tarhan and Yıldırım in 2021 consists of a total of 15 items and 3 sub-dimensions. The Cronbach's alpha internal consistency coefficient of the scale, which has a 5-point Likert-type scoring, was found to be .90 in the total scale and .81 in the professional adaptation sub-dimension; .86 in the communication and cooperation sub-dimension; and .82 in the professional competence sub-dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Beykent University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No